CLINICAL TRIAL: NCT03233867
Title: A Non-interventional Study to Identify Children and Adolescents (Ages 6-17 Years) With Attention Deficit Hyperactivity Disorder and With or Without Copy Number Variants in Specific Genes Involved in Glutamatergic Signaling and Neuronal Connectivity
Brief Title: A Non-interventional Study to Identify Children and Adolescents With ADHD and With or Without mGLuR Mutations
Status: Completed | Type: Observational
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Responsible Party: Sponsor
Organization: Avalo Therapeutics, Inc. (Industry)
Other Study IDs: AEVI-001-ADHD-002
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2018-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional study in children and adolescents (ages 6-17 years) with attention deficit hyperactivity disorder (ADHD) to assess CNVs in specific genes involved in glutamatergic signaling and neuronal connectivity. The screening in this study will be conducted through a combination of online and site performed activities.

ELIGIBILITY:
Inclusion Criteria:

1. Parent/legally authorized representative (LAR) can speak and read English fluently, have provided informed consent and agree to be contacted for an interventional study prior to being genotyped.
2. Subject is 6 to 17 years of age (inclusive) at the time of informed consent.
3. Parent/LAR confirms that the subject has been diagnosed with or been told by a doctor that their child has ADHD.
4. Parent/LAR confirms that the subject is not pregnant and/or breastfeeding.

Exclusion Criteria:

1. Parent/LAR confirms that the subject has been diagnosed with any of the following conditions (aside from ADHD): conduct disorder, anxiety disorder, major depression, autism spectrum disorder (ASD), bipolar disease, psychosis, hypertension, seizure disorder, syncope, or other serious cardiac problems.
2. Aside from your child's current ADHD medication (if applicable), parent/LAR confirms that the subject is currently taking any of the following medications: antidepressants, anti-anxiety medications, anti-psychotics, and/or mood stabilizers.
3. Parent/LAR confirms that the subject has been genotyped previously in the MDGN-NFC1-ADHD-001, MDGN-NFC1-ADHD-101 clinical study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects between the ages of 6 and 17 years, who have been told that they have ADHD, will be eligible for screening.
Sampling Method: Non-Probability Sample
Enrollment: 2503 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Presence of specific copy number variants (CNVs) involved in glutamatergic signaling and neuronal connectivity | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cutler, MD, Principal Investigator — Meridien Research
Locations (1):
- Aevi Genomic Medicine, Wayne, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided